CLINICAL TRIAL: NCT00894322
Title: A Two-Cohort, Single- and Repeat Dose Study to Examine the Pharmacokinetics, Tolerability, and Safety of Ready to Use Exenatide Once Weekly in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Examine the Pharmacokinetics, Tolerability, Safety and Efficacy of Exenatide Once Weekly Suspension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCB110
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Healthy Participants (Experimental): A single 10-mg dose of exenatide once weekly suspension given to healthy participants via 3 subcutaneous (SC) injections at Day 1.
  Interventions: Drug: exenatide once weekly
- Cohort 2: Diabetes Participants (Experimental): On Day 1, participants with type 2 diabetes mellitus treated with diet and exercise alone or with a stable regimen of metformin, thiazolidinedione (TZD), or a combination of metformin or TZD were randomized to receive weekly injections of exenatide suspension for 12 weeks.
  Interventions: Drug: exenatide once weekly
- Cohort 2: Diabetes Participants Placebo (Placebo Comparator): On Day 1, participants with type 2 diabetes mellitus treated with diet and exercise alone or with a stable regimen of metformin, thiazolidinedione (TZD), or a combination of metformin or TZD were randomized to receive weekly injections of medium-chain triglycerides (MCT)-diluent placebo for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 10.0 mg, single injection
  Arms: Cohort 1: Healthy Participants
Drug: exenatide once weekly — subcutaneous injection, 2.0 mg, once a week for 12 weeks
  Arms: Cohort 2: Diabetes Participants
Other: Placebo — subcutaneous injection, volume equivalent to Cohort 2 experimental intervention, once a week for 12 weeks
  Arms: Cohort 2: Diabetes Participants Placebo

SUMMARY:
This study is designed to evaluate the pharmacokinetics, tolerability, and safety of exenatide once weekly suspension in both healthy subjects and in subjects with type 2 diabetes. The study will also evaluate efficacy in the type 2 diabetes patients. Development of this exenatide once weekly presentation would eliminate the need to reconstitute the product prior to use.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Is 19 to 65 years old
* Has a body mass index (BMI) of 23 kg/m2 to 35 kg/m2, inclusive, at study start

Cohort 2:

* Is 19 to 75 years old
* Has been diagnosed with type 2 diabetes mellitus
* Has HbA1c of 7.1% to 10.0%, inclusive, at study start
* Has a body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive, at study start
* Has been treated with diet and exercise alone or with a stable regimen of metformin, a TZD, or a combination of metformin and a TZD, for a minimum of 2 months prior to study start
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to study start:

  * Hormone replacement therapy (female subjects)
  * Oral contraceptives (female subjects)
  * Antihypertensive agents
  * Lipid-lowering agents
  * Thyroid replacement therapy
  * Antidepressant agents

Exclusion Criteria:

Cohort 1:

* Has a personal history of diabetes mellitus (including impaired glucose tolerance, impaired fasting glucose, or gestational diabetes)
* Has received any investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is greater) prior to study start
* Has ever been exposed to exenatide (BYETTA, exenatide once weekly, or any other formulation of exenatide) or any GLP 1 analog

Cohort 2:

* Has received any investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is greater) prior to study start
* Has ever been exposed to exenatide (BYETTA, exenatide once weekly, or any other formulation of exenatide) or any GLP 1 analog
* Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following treatment-excluded medications:

  * Any DPP-4 inhibitor or sulfonylurea (SU) within 3 months prior to study start
  * Alpha glucosidase inhibitor, meglitinide, nateglinide, or pramlintide (SYMLIN®) within 30 days prior to study start
  * Insulin within 2 weeks prior to study start or for more than 1 week within 3 months prior to study start
  * Systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR®) steroids known to have a high rate of systemic absorption
  * Prescription or over-the-counter weight loss medications within 3 months prior to study start

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Amylin Pharmaceuticals, LLC.
Locations (1):
- Research Site, Lincoln, Nebraska, United States

REFERENCES:
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3660&filename=Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants were enrolled in Cohort 1 while participants with type 2 diabetes mellitus were enrolled in Cohort 2.
Pre-assignment Details: Enrolled participants in Cohort 1 were treated on Day 1 only. Enrolled participants who were in Cohort 2 were randomized to one of 2 treatment arms (exenatide or placebo) and were treated for 12 weeks.
Groups:
- Cohort 1 Exenatide 10 mg: A single 10-mg dose of exenatide once weekly suspension was given to healthy participants via 3 subcutaneous (SC) injections at Day 1. At the discretion of the investigator, participants could receive up to 2 anti-emetic medications approximately 30 minutes prior to the exenatide once weekly suspension dose.
- Cohort 2 Exenatide 2 mg: On Day 1, participants with type 2 diabetes mellitus treated with diet and exercise alone or with a stable regimen of metformin, a thiazolidinedione (TZD), or a combination of metformin or a TZD were randomized to receive weekly injections of 2 mg exenatide suspension for 12 weeks. Study medication was administered weekly.
- Cohort 2 Placebo: On Day 1, participants with type 2 diabetes mellitus treated with diet and exercise alone or with a stable regimen of metformin, a thiazolidinedione (TZD), or a combination of metformin or a TZD were randomized to receive weekly injections of medium-chain triglycerides (MCT)-diluent placebo for 12 weeks. Study medication was administered weekly from Visit 2 (Day 1) to Visit 15 (Week 11).
Period: Overall Study
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Started | 30 | 23 | 12
Completed | 29 | 23 | 12
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population. All randomized participants who received at least 1 dose of study medication were included in the ITT population. Totals presented are for only Cohort 2 (35 participants), not for both Cohort 1 and 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo | Total
Number analyzed (Participants) | 30 | 23 | 12 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (14.4) | 52.7 (11.6) | 52.0 (9.3) | 52.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 2 | 23
  Male | 18 | 14 | 10 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 19 | 11 | 53
  Black | 3 | 1 | 0 | 4
  Asian | 0 | 0 | 1 | 1
  Native American | 1 | 1 | 0 | 2
  Hispanic | 3 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 30 | 23 | 12 | 65
Body Weight [Mean (Standard Deviation); unit: kilograms] | 85.9 (15.5) | 104.9 (23.2) | 104.4 (20.3) | 104.7 (22.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was measured in kilograms (kg) of body weight per meter (m) of height, squared.
  kg/m^2 | 28.5 (3.5) | 35.3 (6.7) | 34.9 (4.9) | 35.1 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for Single Dose of 10 mg Exenatide (Cohort 1) in Healthy Participants in the Pharmacokinetic Evaluable Population
Description: Cohort 1: Blood samples for the assessment of plasma exenatide were collected at time = -15, 60, 90, 120, 180, 240, 360, and 480 minutes relative to study medication injection at time = 0 on Day 1 and the mean is presented below. At all visits following the single injection, a single blood sample was collected for assessment of exenatide concentrations. AUC was measured in picograms * hours per milliliter (pg*hr/mL). Exenatide was measured using a validated enzyme-linked immunosorbent assay (ELISA). AUC calculated using linear trapezoidal method from time x to time y; AUC (0-8h) and (0-tlast) are presented below. Pharmacokinetic (PK) evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements [not less than (<) lower limits of quantification (LLOQ)] from Day 1 to Week 12 and had reliable PK data.
Time Frame: Day 1, Week 12
Population: PK evaluable population was analyzed. n in categories below = number of ITT participants with PK evaluable data.
Measure: Geometric Mean (Standard Error); unit: pg*h/mL
Arm/Group | Cohort 1 Exenatide 10 mg
Number analyzed (Participants) | 30
pg*h/mL
  AUC (0-8h), n=30 | 125.6 (41.16)
  AUC (0-Week 12), n=30 | 147220.2 (24000.04)

2. Primary Outcome: Maximum Concentration (Cmax) for Single Dose of 10 mg Exenatide (Cohort 1) in Healthy Participants in the Pharmacokinetic Evaluable Population
Description: Cohort 1: Blood samples for the assessment of plasma exenatide were collected at time = -15, 60, 90, 120, 180, 240, 360, and 480 minutes relative to study medication injection at time = 0 on Day 1 and the mean is presented below. At all visits following the single injection, a single blood sample was collected for assessment of exenatide concentrations. Cmax was measured in picograms per milliliter (pg/mL). Exenatide concentration was measured using a validated enzyme-linked immunosorbent assay (ELISA). PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements [not less than (<) lower limits of quantification (LLOQ)] from Day 1 to Week 12 for the evaluation of the PK characteristics of plasma exenatide and had reliable PK data. Cmax (0-8h) and (0-tlast) are presented below.
Time Frame: Day 1, Week 12
Population: PK evaluable population.
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort 1 Exenatide 10 mg
Number analyzed (Participants) | 30
pg/mL
  Cmax 0 hour to 8 hours | 34.9 (8.33)
  Cmax 0 hour to Week 12 | 331.2 (46.90)

3. Primary Outcome: Time to Maximum Concentration (Tmax) for Single Dose of 10 mg Exenatide (Cohort 1) in Healthy Participants in the Pharmacokinetic Evaluable Population
Description: Cohort 1: Blood samples for the assessment of plasma exenatide were collected at time(t) = -15, 60, 90, 120, 180, 240, 360, and 480 minutes relative to study medication injection at time = 0 on Day 1 an the mean is presented below. At all visits following the single injection, a single blood sample was collected for assessment of exenatide concentrations. Tmax was measured in hours and Tmax (0-8h) and (0-tlast) are presented below. Exenatide concentration was measured using a validated enzyme-linked immunosorbent assay (ELISA). PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements [not less than (<) lower limits of quantification (LLOQ)] and had reliable PK data.
Time Frame: Day 1, Week 12
Population: PK evaluable population. n=number of participants who had reliable PK data available to be evaluated.
Measure: Geometric Mean (Standard Error); unit: hours
Arm/Group | Cohort 1 Exenatide 10 mg
Number analyzed (Participants) | 27
hours
  Tmax (0 to 8 hours), n=27 | 7.0 (0.43)
  Tmax (0 hour to Week 12), n=30 | 998.1 (67.60)

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Injection Site TEAEs, Serious Adverse Events (SAEs), Deaths, and Withdrawals Due to AEs in Cohort 1 and Cohort 2 in Intent to Treat (ITT) Population
Description: Treatment emergent (TE)=occurs during or after treatment with study drug. Adverse Event (AE)=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Participants experiencing multiple episodes of a given AE are counted once. Injection site AEs: adverse events that existed prior to Day 1 and worsened after the first administration at Day 1, or occurred after the first administration at Day 1 through Week 12, or after Study Termination if considered by investigator to be clinically significant.
Time Frame: Day 1 to Week12
Population: ITT population included all participants treated with at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 2 Exenatide 2 mg: On Day 1, participants with type 2 diabetes mellitus treated with diet and exercise alone or with a stable regimen of metformin, a thiazolidinedione (TZD), or a combination of metformin or a TZD were randomized to receive weekly injections of exenatide suspension for 12 weeks. Study medication was administered weekly from Visit 2 (Day 1) to Visit 15 (Week 11).
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 30 | 23 | 12
participants
  TEAE | 26 | 22 | 9
  Injection Site TEAEs | 16 | 18 | 7
  Withdrawal due to AE | 0 | 0 | 0
  SAE | 0 | 0 | 1
  Death | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Concomitant Medications in Cohort 1 and Cohort 2 in ITT Population
Description: Concomitant medications are defined as those medications received on or after the date of the first injection on Day 1, including prior medications that continued past Day 1 and new concomitant medications. Participants may be counted in more than one medication class and no more than once in each class. Categories by Anatomical Therapeutic Chemical (ATC) classification using the World Health Organization (WHO) Drug Dictionary version C1, 01 March 2009. As per protocol, all participants in Cohort 1 could receive up to 2 anti-emetic medications approximately 30 minutes prior to the exenatide.
Time Frame: Day 1 to 12 weeks
Population: ITT population included all participants treated with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 30 | 23 | 12
participants | 30 | 21 | 11

6. Secondary Outcome: AUC (0 Hour to 168 Hour) for 10 mg Exenatide (Cohort 1) in Healthy Participants in the Pharmacokinetic Evaluable Population
Description: Cohort 1: Blood samples for the assessment of plasma exenatide were collected at time = -15, 60, 90, 120, 180, 240, 360, and 480 minutes relative to study medication injection at time = 0 on Day 1. At all visits following the single injection, a single blood sample was collected for assessment of exenatide concentrations. AUC (0-168 h) data represents average concentration rather than maximum concentration. Exenatide concentration was measured using a validated enzyme-linked immunosorbent assay (ELISA). AUC calculated using linear trapezoidal method from time x to time y and measured in pg*h/mL. PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements (not < LLOQ) from Day 1 to Week 12 and had reliable PK data.
Time Frame: Day 1 to Week 1
Population: PK evaluable population.
Measure: Geometric Mean (Standard Error); unit: pg*h/mL
Arm/Group | Cohort 1 Exenatide 10 mg
Number analyzed (Participants) | 30
pg*h/mL | 3269.6 (1661.45)

7. Secondary Outcome: Average Exenatide Concentration (Cave) of 10 mg Exenatide (Cohort 1) in Healthy Participants in the Pharmacokinetic Evaluable Population
Description: Cohort 1: Blood samples for the assessment of plasma exenatide were collected at time = -15, 60, 90, 120, 180, 240, 360, and 480 minutes relative to study medication injection at time = 0 on Day 1. At all visits following the single dose, a single blood sample was collected for assessment of exenatide concentrations. Cave(0-168h) was the time-weighted mean concentration over the sampling period from time x to time y corresponding to AUC (0-168h) and was measured in picograms per milliliter (pg/mL). Exenatide concentration was measured using a validated enzyme-linked immunosorbent assay (ELISA). PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements [not less than (<) lower limits of quantification (LLOQ)] from Day 1 to Week 12 and had reliable PK data.
Time Frame: Day 1 to Week 1
Population: PK evaluable population.
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort 1 Exenatide 10 mg
Number analyzed (Participants) | 30
pg/mL | 32.5 (7.53)

8. Primary Outcome: Mean Change From Baseline to End of Study in Sitting Diastolic and Systolic Blood Pressure in Cohorts 1 and 2 in ITT Population
Description: In Cohort 1, sitting blood pressures were obtained at Screening (Visit 1), Day 1 (Visit 2), Weeks 1-11 (Visits 3-13), Week 12 (Visit 14), and at early termination. Blood pressures (diastolic and systolic) were measured in millimeters of mercury (mmHg). In Cohort 2, sitting blood pressures were obtained at Screening (Visit 1), Day 1 (Visit 2), Weeks 1-10 (Visits 3-12), Week 11 (Visit 15), Week 12 (Visit 16) and at early termination. Baseline was defined as last measurement prior to first injection of study drug.
Time Frame: Day 1 to Week 12
Population: ITT population included all participants treated with at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 30 | 23 | 12
mmHg
  Diastolic Blood Pressure | 6.2 (7.05) | 4.6 (8.81) | 6.8 (7.81)
  Systolic Blood Pressure | -1.4 (9.59) | -8.4 (14.15) | -1.7 (12.47)

9. Primary Outcome: Mean Change From Baseline to End of Study in Sitting Heart Rate in Cohorts 1 and 2 in ITT Population
Description: In Cohort 1, sitting heart rates were obtained at Screening (Visit 1), Day 1 (Visit 2), Weeks 1-11 (Visits 3-13), Week 12 (Visit 14), and at early termination. Heart rate was measured in beats per minute (bpm). In Cohort 2, sitting heart rates were obtained at Screening (Visit 1), Day 1 (Visit 2), Weeks 1-10 (Visits 3-12), Week 11 (Visit 15), Week 12 (Visit 16) and at early termination. Baseline was defined as last measurement prior to first injection of study drug.
Time Frame: Day 1 to Week 12
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 30 | 23 | 12
bpm | -7.5 (9.38) | -5.4 (8.10) | -9.1 (7.03)

10. Primary Outcome: Number of Participants With Hematology and Serum Chemistry Laboratory Values of Potential Clinical Importance in Cohorts 1 and 2 in ITT Population
Description: Abbreviations: Upper Limit of Normal (ULN); milligram per deciliter (mg/dL); units per liter (U/L); micro liters (µL); creatine kinase (CK); gamma-glutamyltransferase (G-GT). Normal ranges = Hematocrit: 40.6-52.3% (male), 35.3-47.0 (female); Platelets 155-361*10^3/µL(male/female); Calcium: 8.6-10.4 mg/dL (male/female); CK: 43-350 U/L (male), 28-207 U/L (female); G-GT: 7-62 U/L (male/female); Glucose 73-105 mg/dL (male/female); Lipase 14-70 U/L (male/female); Uric acid: 3.5-7.8 mg/dL (male), 2.3-5.9 mg/dL (female). Blood samples for laboratories were collected at screening, Day 1, Weeks 4, 8, 12 or early termination. Value for potential clinical importance is presented in each category presented below.
Time Frame: Day 1 to Week 12
Population: ITT population included all participants treated with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 30 | 23 | 12
participants
  Hematocrit low <36% | 0 | 0 | 1
  Platelets high <75 to >500*10^3/µ/L | 0 | 1 | 0
  Calcium high <8 to >11 mg/dL | 0 | 1 | 0
  CK high >3*ULN | 1 | 0 | 0
  G-GT high >3*ULN in U/L | 0 | 0 | 1
  Glucose low <50 to > 450 mg/dL | 1 | 0 | 0
  Lipase high >3*ULN in U/L | 0 | 0 | 1
  Uric Acid high >8.0 mg/dL | 0 | 1 | 0

11. Primary Outcome: Antibody Titers for Participants With Treatment Emergent Positive Antibodies to Exenatide in Participants Who Received Exenatide in Cohorts 1 and 2
Description: Serum titers of antibodies to exenatide were evaluated using a validated enzyme-linked immunosorbent assay (Covance Method No. ELISA-0308). Positive antibody to exenatide titer: observed at the indicated visit following a negative or missing titer at baseline, or a positive titer that has increased by at least 3 dilutions at the indicated visit from a detectable baseline. Baseline=Day 1. Negative titers were assigned a value of 1 in order to calculate geometric mean. Geometric mean of reportable titers, by study week, are presented below.
Time Frame: Day 1 to Week 12
Population: Only participants who received exenatide were analyzed (no placebo-treated participants were included). N=number of participants in each treatment at each visit and n= number of participants with reportable titers at the visit. Last visit=last visit with reportable titers.
Measure: Geometric Mean (Standard Error); unit: Reportable Titers
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg
Number analyzed (Participants) | 30 | 23
Reportable Titers
  Week 2, N=30, 23; n=4, 1 | 25.0 (0.0) | 25.0 (NA) — Only 1 participant with reportable titer so SE cannot be calculated.
  Week 4, N=30, 23; n=14, 10 | 394.6 (204.4) | 202.6 (109.2)
  Week 6, N=30, 23; n=0, 15 | NA (NA) — No reportable titers (n=0) available for this week in this treatment group so mean (SE) are not applicable (n/a) | 295.9 (129.9)
  Week 8, N=29, 23; n=22,15 | 300.7 (118.0) | 561.4 (186.4)
  Week 10, N=29, 23; n=0,15 | NA (NA) — No reportable titers (n=0) available for this week in this treatment group so mean (SE) are not applicable (n/a) | 453.0 (190.9)
  Last visit, N=30, 23; n=20, 15 | 202.6 (63.0) | 625.0 (294.5)

12. Secondary Outcome: Least Square Mean Change From Baseline in Hemoglobin A1c (HbA1c) to Week 12 in Participants With Diabetes (Cohort 2) in the ITT Population
Description: HbA1c was measured as a percent of hemoglobin at screening, Day 1, Weeks 4, 8, 12 or early termination. Last observation carried forward (LOCF) was applied to estimate missing values at post baseline timepoints. Baseline=Day 1, last measurement prior to first dose of study drug.
Time Frame: Day 1 to Week 12
Population: ITT population included all participants treated with at least one dose of study drug. This analysis was only done in Cohort 2 so the ITT population of Cohort 2 was available for analysis.
Measure: Least Squares Mean (Standard Error); unit: Percent of hemoglobin
Arm/Group | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 23 | 12
Percent of hemoglobin | -0.87 (0.179) | 0.08 (0.231)
Statistical Analysis 1: Comparison: Cohort 2 Exenatide 2 mg vs Cohort 2 Placebo; Test type: Superiority or Other; p = 0.0013, ANOVA — Treatment group and HbA1c stratum at screening were factors. Placebo was reference group; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.50 to -0.40], Standard Error of Mean 0.269

13. Secondary Outcome: Number of Participants Achieving HbA1c Less Than Equal to (<=) 6.5% and Less Than (<) 7% at Week 12 in Participants With Diabetes (Cohort 2) in the ITT Population
Description: HbA1c was measured as a percent of hemoglobin at screening, Day 1, Weeks 4, 8, 12 or early termination. LOCF was applied to estimate missing values at post baseline timepoints. Baseline=Day 1, last measurement prior to first dose of study drug.
Time Frame: Week 12
Population: ITT population included all participants treated with at least one dose of study drug. Only those ITT participants in Cohort 2 were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 23 | 12
participants
  Baseline HbA1c >= 7% | 22 | 12
  Week 12 HbA1c <= 6.5% | 9 | 1
  Week 12 HbA1c <7% | 14 | 2
Statistical Analysis 1: Comparison: Cohort 2 Exenatide 2 mg vs Cohort 2 Placebo; Test type: Superiority or Other; p = 0.0033, Cochran-Mantel-Haenszel; Adjusted for HbA1c strata at screening

14. Secondary Outcome: Mean Change From Baseline at Week 12 in Body Weight in Participants With Diabetes (Cohort 2) in the ITT Population
Description: Body weight was measured in kilograms (kg). Baseline was Day 1, last measurement prior to first dose of study drug. Body weight was measured at screening, Day 1, Weeks 4, 8, 12 or early termination and the LOCF approach was applied to estimate missing value at each post baseline timepoint.
Time Frame: Baseline, Week 12
Population: ITT population included all participants treated with at least one dose of study drug. Only Cohort 2 was analyzed for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 23 | 12
kg | -1.41 (0.558) | -0.39 (0.717)
Statistical Analysis 1: Comparison: Cohort 2 Exenatide 2 mg vs Cohort 2 Placebo; Least square mean (LS) mean, 95% confidence interval (CI) and p-value calculated for the changes in weight from baseline in participants in cohort 2 treated with exenatide with placebo as reference group; Test type: Superiority or Other; p = 0.2285, ANOVA; treatment group and HbA1c stratum at screening were factors; LS Mean Difference = -1.03, 95% CI 2-sided [-2.73 to 0.68], Standard Error of Mean 0.835

15. Secondary Outcome: Mean Change From Baseline at Week 12 in Fasting Plasma Glucose in Participants With Diabetes (Cohort 2) for the ITT Population
Description: Baseline was the last measurement at the screening visit. Fasting plasma glucose (FPG) was measured at screening, Day 1, Weeks 2, 4, 6, 8, 12, or early termination and reported in milligrams per deciliter (mg/dL).
Time Frame: Baseline, Week 12
Population: ITT population included all participants treated with at least one dose of study drug. Only participants in Cohort 2 were evaluated for this Outcome Measure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Number analyzed (Participants) | 23 | 12
mg/dL | -32 (9.9) | 8 (11.9)
Statistical Analysis 1: Comparison: Cohort 2 Exenatide 2 mg vs Cohort 2 Placebo; Test type: Superiority or Other; p = 0.0035, ANOVA; treatment group and HbA1c stratum at screening were factors; LS Mean Difference = -40.4, 95% CI 2-sided [-66.5 to -14.3], Standard Error of Mean 12.8

16. Primary Outcome: Area Under the Curve (AUC) for 2 mg Exenatide (Cohort 2) in Participants With Diabetes in the Pharmacokinetic Evaluable Population
Description: Cohort 2: Blood samples for the assessment of plasma exenatide were collected on Day 1, Weeks 2, 4, 6, 8, and 10. At Week 10, blood samples were collected at time = -15, 60, 90, 120, 180, 240, and 360 minutes relative to study medication injection at time = 0. AUC was measured in picograms * hours per milliliter (pg*hr/mL). Exenatide was measured using a validated enzyme-linked immunosorbent assay (ELISA). AUC calculated using linear trapezoidal method from time x to time y; AUC (0-6h) measured at Week 10, AUC (0-168h) steady state measured between Weeks 10 and 11, and AUC (0-tlast) for time interval between Weeks 10 and 12 (approximately336 hours) are presented below. PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements (not < LLOQ) from Day 1 to Week 12 and had reliable PK data.
Time Frame: Week 10-11; Weeks 10 - 12
Population: PK evaluable population was analyzed. In categories below, n = number of ITT participants with PK evaluable data. Note: Placebo-treated participants not included in this analysis.
Measure: Geometric Mean (Standard Error); unit: pg*hr/mL
Arm/Group | Cohort 2 Exenatide 2 mg
Number analyzed (Participants) | 18
pg*hr/mL
  AUC (0-6h) at Week 10, n=18 | 1535.3 (232.40)
  AUC (0-168h) at Weeks 10-11, n=18 | 49100.2 (6796.56)
  AUC (0-tlast) at Weeks 10-12, n=17 | 101615.0 (12927.42)

17. Primary Outcome: Average Exenatide Concentration (Cave) of 2 mg Exenatide (Cohort 2) in Participants With Diabetes in the Pharmacokinetic Evaluable Population
Description: Cohort 2: Blood samples for the assessment of plasma exenatide were collected on Day 1, Weeks 2, 4, 6, 8, and 10. At Week 10, blood samples were collected at time = -15, 60, 90, 120, 180, 240, and 360 minutes relative to study medication injection at time = 0. At all visits following the single injection, a single blood sample was collected for assessment of exenatide concentrations. Cave(0-168h) and Cave(0-tlast) was the time-weighted mean concentration over the sampling period from time x to time y corresponding to AUC (0-168h), and AUC (0-tlast), respectively. Cave was measured in picograms per milliliter (pg/mL). Exenatide concentration was measured using a validated enzyme-linked immunosorbent assay (ELISA). PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements (not < LLOQ) from Day 1 to Week 12 and had reliable PK data.
Time Frame: Week 10 - Week 11; Week 10 - Week 12
Population: as for outcome 16
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort 2 Exenatide 2 mg
Number analyzed (Participants) | 18
pg/mL
  Cave at Weeks 10-11; n=18 | 292.7 (40.52)
  Cave at Weeks 10-12; n=17 | 302.4 (38.47)

18. Primary Outcome: Maximum Concentration (Cmax) for 2 mg Exenatide (Cohort 2) in Participants With Diabetes in the Pharmacokinetic Evaluable Population
Description: Cohort 2: Blood samples for the assessment of plasma exenatide were collected on Day 1, Weeks 2, 4, 6, 8, and 10. At Week 10, blood samples were collected at time = -15, 60, 90, 120, 180, 240, and 360 minutes relative to study medication injection at time = 0. Cmax was measured in pg/mL. Exenatide was measured using a validated enzyme-linked immunosorbent assay (ELISA). Cmax summarized at 0-6 h at Week 10, 0-168 h at Weeks 10-11, and 0-tlast at Weeks 10-12. PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements (not < LLOQ) from Day 1 to Week 12 and had reliable PK data.
Time Frame: Week 10, Weeks 10-11, Weeks 10-12
Population: as for outcome 16
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Cohort 2 Exenatide 2 mg
Number analyzed (Participants) | 18
pg/mL
  Cmax at 0-6 h Week 10; n=18 | 304.9 (47.39)
  Cmax at 0-168 h Weeks 10=11; n=18 | 362.6 (50.86)
  Cmax at 0-tlast Weeks 10-12; n=17 | 410.5 (53.27)

19. Primary Outcome: Time to Maximum Concentration (Tmax) of 2 mg Exenatide (Cohort 2) in Participants With Diabetes in Pharmacokinetic Evaluable Population
Description: Cohort 2: Blood samples for the assessment of plasma exenatide were collected on Day 1, Weeks 2, 4, 6, 8, and 10. At Week 10, blood samples were collected at time = -15, 60, 90, 120, 180, 240, and 360 minutes relative to study medication injection at time = 0. Tmax was measured in hours (h). Exenatide was measured using a validated ELISA. Tmax summarized at 0-6 h at Week 10, 0-168 h at Weeks 10-11, and 0-tlast at Weeks 10-12. PK evaluable population consisted of all ITT participants who had at least 4 detectable plasma exenatide measurements (not < LLOQ) from Day 1 to Week 12 and had reliable PK data.
Time Frame: Week 10, Weeks 10-11, Weeks 10-12
Population: as for outcome 16
Measure: Geometric Mean (Standard Error); unit: hours
Arm/Group | Cohort 2 Exenatide 2 mg
Number analyzed (Participants) | 18
hours
  Tmax 0-6 h Week; n=18 | 1.4 (0.20)
  Tmax 0-168 h Weeks 10-11; n=18 | 34.3 (13.96)
  Tmax 0-tlast Weeks 10-12; n=17 | 60.0 (26.01)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Arm/Group | Cohort 1 Exenatide 10 mg | Cohort 2 Exenatide 2 mg | Cohort 2 Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/23 | 1/12
Other Adverse Events (participants affected / at risk) | 26/30 | 22/23 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Exenatide 10 mg (N=30) | Cohort 2 Exenatide 2 mg (N=23) | Cohort 2 Placebo (N=12)
Infected Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Exenatide 10 mg (N=30) | Cohort 2 Exenatide 2 mg (N=23) | Cohort 2 Placebo (N=12)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
Feeling hot (General disorders) | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 1 | 0
Infection site erythema (General disorders) | 4 | 12 | 1
Injection site hematoma (General disorders) | 5 | 9 | 6
Injection site pain (General disorders) | 6 | 5 | 0
Injection site papule (General disorders) | 1 | 0 | 0
Injection site pruritus (General disorders) | 10 | 11 | 1
Injection site swelling (General disorders) | 1 | 0 | 0
Injection site warmth (General disorders) | 0 | 2 | 0
Edema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Vessel puncture site hematoma (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blister (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 6 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.